CLINICAL TRIAL: NCT05649917
Title: A Post-Market Observational Case Series Study of Percutaneous Peripheral Nerve Stimulation (PNS) for the Treatment of Chronic Shoulder Pain
Brief Title: SPR PNS for Chronic Shoulder Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: International Spine, Pain and Performance Center (Other)
Collaborators: SPR Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Mehul J. Desai, Study Principal Investigator, International Spine, Pain and Performance Center
Other Study IDs: 20223406
Record Dates: First submitted 2022-08-23; First posted 2022-12-14 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Shoulder Pain; Shoulder Injuries; Shoulder Arthritis
Keywords: Peripheral Nerve Stimulation; Shoulder Pain; Shoulder Injuries
MeSH Terms: conditions — Shoulder Pain; Shoulder Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this research is to gather post-market data regarding the effectiveness of the SPRINT Peripheral Nerve Stimulation (PNS) System for the treatment of chronic shoulder pain due to chronic degenerative changes of your shoulder. The System delivers mild electrical stimulation to the muscles in your shoulder. The System includes up to two leads (small wires) that are placed through your skin into your shoulder. The leads attach to a device worn on your body that deliver stimulation (called a Stimulator). The device is cleared by the FDA for up to 60 days of use for the relief of chronic or acute pain.

DETAILED DESCRIPTION:
Background

Chronic degenerative changes in the shoulder are a frequent source of debilitating chronic pain. In particular, osteoarthritis of the shoulder has been estimated to affect up to 32.8% of the adult population over the age of 60, and OA in general is one of the most frequent causes of disability in the United States.1 OA impacts the quality of life of tens of millions of Americans and carries a significant economic burden of over $60 billion in the U.S. each year.2

Degenerative joint disease in the shoulder is commonly managed with physical therapy and over-the-counter medications, but these modalities can be insufficient for pain management as degeneration progresses.3 Corticosteroid injections, radiofrequency ablations, and even partial or total shoulder arthroplasty are used to treat advanced cases3, and these interventions often either have limited long-term effectiveness or are associated with significant invasiveness or other side effects and complications.

Peripheral nerve stimulation (PNS) is a neuromodulatory technique that seeks to provide pain relief through stimulation of the nerves that innervate the shoulder (e.g., the suprascapular nerve and axillary nerve). A novel, 60-day percutaneous PNS system that is FDA-cleared has shown effectiveness for chronic shoulder pain following stroke and shoulder impingement syndrome4-15, and has demonstrated the potential to provide sustained relief following the short-term, 60-day treatment.8, 15-18 The mechanism of action of neuropathic pain in osteoarthritis is proposed to be via peripheral sensitization (e.g., axillary and suprascapular nerves) that leads to subsequent upstream hypersensitization of the central nervous system; the proposed mechanism of long-term pain relief with 60-day PNS via reconditioning of the CNS to reverse hypersensitization therefore suggests that the treatment may be effective for degenerative shoulder including OA.19, 20 However, no study has prospectively evaluated the use of 60-day, percutaneous PNS for the treatment of debilitating pain associated with degenerative changes in the shoulder. The goal of this study is therefore to collect data on the use of 60-day PNS for the treatment of chronic pain associated with degenerative shoulder.

Objectives

The study objective is to gather post-market data regarding the effectiveness of the SPRINT PNS System for the treatment of chronic shoulder pain due to degenerative changes of the shoulder.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years old
* Diagnosed with degenerative changes within the shoulder complex
* Scheduled for a commercial SPRINT PNS procedure
* Shoulder pain score at baseline >5 as demonstrated by PROMIS 29
* Able to understand and willing to take part in study and comply with all study requirements

Exclusion Criteria:

* No shoulder pain at rest
* Pain exclusively in the anterior aspect of the shoulder
* Confounding conditions such as cervical radiculopathy, inflammatory arthritis, complete rotator cuff tear, or ipsilateral shoulder surgery in the past one year
* Daily opioid use >90 m morphine equivalent at any point in the past month
* Opioids for any condition other than shoulder pain
* Deep brain stimulation (DBS) system, implanted active cardiac implant (e.g. pacemaker or defibrillator), or any other implantable neuro-stimulator whose stimulus current pathway may overlap with the SPRINT system.
* Any other condition that may interfere with the ability to participate in a clinical trial (e.g. anatomy that may interfere with lead placement, nerve damage, compromised immune system, uncontrolled DM) as determined by the Investigator
* Vulnerable populations (e.g., prisoners, minors, students, employees)
* Workers Compensation
* Pregnant

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will enroll up to 20 patients with pain due to degenerative changes in the shoulder scheduled for commercial placement of the SPRINT PNS System.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Reduction in average pain and/or reduction in pain interference | 3 months
  Average pain intensity is measured using the PROMIS-29 v2.0 profile. The measure assesses pain intensity using a single 0-10 numeric rating scale. Average pain interference is measured using Brief Pain Inventory--Short Form Question #9 (BPI-9). BPI-9 uses a 0-10 numeric rating scale across seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance.)

SECONDARY OUTCOMES:
Changes in pain intensity | 1 year
  Changes in pain intensity will be assessed using the PROMIS-29 v2.0 profile. The measure assesses pain intensity using a single 0-10 numeric rating scale.
Changes in pain interference | 1 year
  Changes in average pain interference are measured using Brief Pain Inventory--Short Form Question #9. The measure assesses pain interference using a 0-10 numeric rating scale across seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance.)
Changes in Shoulder Function | 1 year
  Shoulder function is measured using the Western Ontario Arthritis of the Shoulder (WOOS) index. The WOOS index is a patient-reported, disease-specific questionnaire for the measurement of the quality-of-life in patients with osteoarthritis.
Changes in shoulder range of motion | 1 year
  Shoulder range of motion is measured as degrees of active range of motion (flexion, abduction, internal rotation, and external rotation) based on physical examination.

CONTACTS AND LOCATIONS:
Overall Officials: Mehul Desai, MD, MPH, Principal Investigator — International Spine Pain & Performance Center
Locations (2):
- United States (2):
  - International Spine Pain & Performance Center, Washington D.C., District of Columbia
  - International Spine Pain & Performance Center, Arlington, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chillemi C, Franceschini V. Shoulder osteoarthritis. Arthritis. 2013;2013:370231. doi: 10.1155/2013/370231. Epub 2013 Jan 10. PMID 23365745
- [Background] Buckwalter JA, Saltzman C, Brown T. The impact of osteoarthritis: implications for research. Clin Orthop Relat Res. 2004 Oct;(427 Suppl):S6-15. doi: 10.1097/01.blo.0000143938.30681.9d. PMID 15480076
- [Background] Millett PJ, Gobezie R, Boykin RE. Shoulder osteoarthritis: diagnosis and management. Am Fam Physician. 2008 Sep 1;78(5):605-11. PMID 18788237
- [Background] Chae J, Yu D, Walker M. Percutaneous, intramuscular neuromuscular electrical stimulation for the treatment of shoulder subluxation and pain in chronic hemiplegia: a case report. Am J Phys Med Rehabil. 2001 Apr;80(4):296-301. doi: 10.1097/00002060-200104000-00014. PMID 11277137
- [Background] Yu DT, Chae J, Walker ME, Fang ZP. Percutaneous intramuscular neuromuscular electric stimulation for the treatment of shoulder subluxation and pain in patients with chronic hemiplegia: a pilot study. Arch Phys Med Rehabil. 2001 Jan;82(1):20-5. doi: 10.1053/apmr.2001.18666. PMID 11239281
- [Background] Renzenbrink GJ, IJzerman MJ. Percutaneous neuromuscular electrical stimulation (P-NMES) for treating shoulder pain in chronic hemiplegia. Effects on shoulder pain and quality of life. Clin Rehabil. 2004 Jun;18(4):359-65. doi: 10.1191/0269215504cr759oa. PMID 15180118
- [Background] Yu DT, Chae J, Walker ME, Kirsteins A, Elovic EP, Flanagan SR, Harvey RL, Zorowitz RD, Frost FS, Grill JH, Feldstein M, Fang ZP. Intramuscular neuromuscular electric stimulation for poststroke shoulder pain: a multicenter randomized clinical trial. Arch Phys Med Rehabil. 2004 May;85(5):695-704. doi: 10.1016/j.apmr.2003.07.015. PMID 15129391
- [Background] Chae J, Yu DT, Walker ME, Kirsteins A, Elovic EP, Flanagan SR, Harvey RL, Zorowitz RD, Frost FS, Grill JH, Fang ZP. Intramuscular electrical stimulation for hemiplegic shoulder pain: a 12-month follow-up of a multiple-center, randomized clinical trial. Am J Phys Med Rehabil. 2005 Nov;84(11):832-42. doi: 10.1097/01.phm.0000184154.01880.72. PMID 16244520
- [Background] Chae J, Ng A, Yu DT, Kirsteins A, Elovic EP, Flanagan SR, Harvey RL, Zorowitz RD, Fang ZP. Intramuscular electrical stimulation for shoulder pain in hemiplegia: does time from stroke onset predict treatment success? Neurorehabil Neural Repair. 2007 Nov-Dec;21(6):561-7. doi: 10.1177/1545968306298412. Epub 2007 Mar 16. PMID 17369520
- [Background] Wilson RD, Bennett ME, Lechman TE, Stager KW, Chae J. Single-lead percutaneous peripheral nerve stimulation for the treatment of hemiplegic shoulder pain: a case report. Arch Phys Med Rehabil. 2011 May;92(5):837-40. doi: 10.1016/j.apmr.2010.11.003. PMID 21530732
- [Background] Wilson RD, Harris MA, Bennett ME, Chae J. Single-lead percutaneous peripheral nerve stimulation for the treatment of shoulder pain from subacromial impingement syndrome. PM R. 2012 Aug;4(8):624-8. doi: 10.1016/j.pmrj.2012.03.002. PMID 22920317
- [Background] Chae J, Wilson RD, Bennett ME, Lechman TE, Stager KW. Single-lead percutaneous peripheral nerve stimulation for the treatment of hemiplegic shoulder pain: a case series. Pain Pract. 2013 Jan;13(1):59-67. doi: 10.1111/j.1533-2500.2012.00541.x. Epub 2012 Mar 26. PMID 22448759
- [Background] Wilson RD, Gunzler DD, Bennett ME, Chae J. Peripheral nerve stimulation compared with usual care for pain relief of hemiplegic shoulder pain: a randomized controlled trial. Am J Phys Med Rehabil. 2014 Jan;93(1):17-28. doi: 10.1097/PHM.0000000000000011. PMID 24355994
- [Background] Wilson RD, Harris MA, Gunzler DD, Bennett ME, Chae J. Percutaneous peripheral nerve stimulation for chronic pain in subacromial impingement syndrome: a case series. Neuromodulation. 2014 Dec;17(8):771-6; discussion 776. doi: 10.1111/ner.12152. Epub 2014 Feb 11. PMID 24512114
- [Background] Wilson RD, Bennett ME, Nguyen VQC, Bock WC, O'Dell MW, Watanabe TK, Amundson RH, Hoyen HA, Chae J. Fully Implantable Peripheral Nerve Stimulation for Hemiplegic Shoulder Pain: A Multi-Site Case Series With Two-Year Follow-Up. Neuromodulation. 2018 Apr;21(3):290-295. doi: 10.1111/ner.12726. Epub 2017 Nov 22. PMID 29164745
- [Background] Gilmore CA, Ilfeld BM, Rosenow JM, Li S, Desai MJ, Hunter CW, Rauck RL, Nader A, Mak J, Cohen SP, Crosby ND, Boggs JW. Percutaneous 60-day peripheral nerve stimulation implant provides sustained relief of chronic pain following amputation: 12-month follow-up of a randomized, double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2019 Nov 17:rapm-2019-100937. doi: 10.1136/rapm-2019-100937. Online ahead of print. PMID 31740443
- [Background] Gilmore CA, Kapural L, McGee MJ, Boggs JW. Percutaneous Peripheral Nerve Stimulation for Chronic Low Back Pain: Prospective Case Series With 1 Year of Sustained Relief Following Short-Term Implant. Pain Pract. 2020 Mar;20(3):310-320. doi: 10.1111/papr.12856. Epub 2019 Dec 2. PMID 31693791
- [Background] Mainkar O, Solla CA, Chen G, Legler A, Gulati A. Pilot Study in Temporary Peripheral Nerve Stimulation in Oncologic Pain. Neuromodulation. 2020 Aug;23(6):819-826. doi: 10.1111/ner.13139. Epub 2020 Mar 17. PMID 32185844
- [Background] Deer TR, Eldabe S, Falowski SM, Huntoon MA, Staats PS, Cassar IR, Crosby ND, Boggs JW. Peripherally Induced Reconditioning of the Central Nervous System: A Proposed Mechanistic Theory for Sustained Relief of Chronic Pain with Percutaneous Peripheral Nerve Stimulation. J Pain Res. 2021 Mar 12;14:721-736. doi: 10.2147/JPR.S297091. eCollection 2021. PMID 33737830
- [Background] Dimitroulas T, Duarte RV, Behura A, Kitas GD, Raphael JH. Neuropathic pain in osteoarthritis: a review of pathophysiological mechanisms and implications for treatment. Semin Arthritis Rheum. 2014 Oct;44(2):145-54. doi: 10.1016/j.semarthrit.2014.05.011. Epub 2014 May 14. PMID 24928208